CLINICAL TRIAL: NCT01390870
Title: Establishing Predictors of Enlarged Prostate Treatment Adherence: Linking Symptom Improvement to Adherence
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112597
Record Dates: First submitted 2011-04-14; First posted 2011-07-11 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia
Keywords: Enlarged prostate, 5-alpha-reductase inhibitor, alpha-blocker, adherence
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Survey: Men from the United States aged 50 years or older who initiated medication for EP within the past 12 months.
  Interventions: Drug: 5ARI or AB or Combination Therapy (5ARI + AB)

INTERVENTIONS:
Drug: 5ARI or AB or Combination Therapy (5ARI + AB) — 5ARI: Dutasteride or Finasteride; AB: Doxazosin, Silodosin, Tamsulosin, Terazosin, or Alfuzosin
  Other Names: Hytrin® is a registered trademark of Abbott Labs; Uroxatral® is a registered trademark of Sanofi-Aventis; Avodart® is a registered trademark of GlaxoSmithKline; Cardura® is a registered trademark of Pfizer; Rapaflo® is a registered trademark of Watson Pharma Inc; Proscar® is a registered trademark of Merck; Flomax® is a registered trademark of Boehringer-Ingelheim

SUMMARY:
Patient-based surveys will be conducted to evaluate the drivers of medication adherence in patients treated with either 5-alpha-reductase inhibitor (5ARI) therapy, alpha-blocker (AB) therapy, or combination therapy for enlarged prostate (EP). Adherence with EP therapy will be evaluated. The researchers believe that the majority of participants will report that they are compliant with therapy. The data source is a cross-sectional patient survey administered at one time point.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged 50 years or older
* Residents of the United States
* Receiving a prescription for an enlarged prostate (EP) treatment within 12 months prior to survey initiation

Exclusion Criteria:

* Patients with prostate cancer
* no health/prescription insurance
* patients receiving medication(s) for EP on a PRN basis

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  * Physician confirmed diagnosis of enlarged prostate (EP)
  * Age 50 or older
  * Resident of the United States with health insurance that covers prescription drugs
  * EP is consistently treated with a medication that was intiated within the previous 12 months
  Exclusion criteria
  * age less than 50
  * receiving medication on an as needed basis
  * diagnosis of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a participant cohort. All diagnoses and treatment are recorded in the course of routine medical practice.
Groups:
- All Enrolled Participants: Males at least 50 years of age who were residents of the United States with one or more diagnoses of enlarged prostate and one or more filled prescription medications within the past 12 months for enlarged prostate (EP) (alpha blocker [AB], 5-alpha reductase inhibitor [5-ARI], combination therapy)
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 400
Completed | 400
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 400
Age, Customized [Number; unit: Participants] — The number of participants who were aged 50 and older and those aged 49 and younger are presented.
  Participants
    at least 50 years old | 400
    less than 50 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 400
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 391
  African American | 2
  Hispanic | 1
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Compliance With Medication
Description: Compliance was calculated based on the participant's response to the following question: "In general, how many times did you miss taking your prostate medication?" Responses were measured on a 5-point scale. Participants who answered "I never miss a dose of my medication" were considered compliant. All other responses were considered non-compliant.
Time Frame: Cross sectional survey administered once to each participant during a 17-month study period (May 2009 to September 2010)
Population: All enrolled participants taking 5-alpha reductase inhibitors and/or alpha blockers
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 400
participants
  Compliant | 239
  Non-Compliant | 161

ADVERSE EVENTS:
Description: This was a survey of participants, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.